CLINICAL TRIAL: NCT00849108
Title: A Phase 2, Open-Label, Randomized Multicenter Study for the Development of One-Day Rest/Stress Cardiac Positron Emission Tomography (PET) Perfusion Imaging Protocols of BMS747158
Brief Title: Development of 1-Day Rest/Stress Cardiac PET Perfusion Imaging Protocol of BMS747158
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BMS747158-201
Record Dates: First submitted 2009-01-05; First posted 2009-02-23 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2012-04

CONDITIONS: Ischemia
Keywords: Myocardial Perfusion; PET imaging; SPECT imaging; Coronary artery disease; Subjects that are male and nonpregnant female patients; presenting with reversible ischemia as characterized by a; rest/stress SPECT imaging study using; Technetium(99mTc)-labeled tracers
MeSH Terms: conditions — Ischemia; Coronary Artery Disease | interventions — BMS 747158-02

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1: dose range and dose interval (Experimental): Patients to receive either 2 or 3 IV bolus injections of BMS747158: 1 at rest and 1 or 2 during pharmacological or exercise stress, over a 1-day or 2-day period.
  Interventions: Drug: BMS747158
- Cohort 2: Pharm&exercise stress Efficacy (Experimental): Patients to receive 2 IV bolus injections of BMS747158:1 at rest and 1 at stress
  For the Pharmacologic (Adenosine) Stress:
  * Doses at rest to range between 2.9 and 3.4 mCi.
  * Doses under stress to be a factor of 2.0 to 2.4 greater than the rest dose, resulting in a range of stress doses between 5.8 and 8.2 mCi.
  For the Exercise Stress:
  * Doses at rest were to range between 1.7 and 2.0 mCi.
  * Doses under stress were to be a factor of 3.0 to 3.6 greater than the rest dose, resulting in a range between 5.1 and 7.2 mCi.
  Interventions: Drug: BMS747158

INTERVENTIONS:
Drug: BMS747158 — dosages at rest and at stress were not to exceed a total of 14 mCi.
  Cohort 1: Patients received either 2 or 3 IV bolus injections of BMS747158: 1 at rest and 1 or 2 during stress, over a 1-day or 2-day period.
  Cohort 2: Patients to recieve IV bolus injections of BMS747158:
  For the Pharmacologic (Adenosine) Stress:
  * Doses at rest were to range between 2.9 and 3.4 mCi.
  * Doses under stress were to be a factor of 2.0 to 2.4 greater than the rest dose, resulting in a range of stress doses between 5.8 and 8.2 mCi.
  For the Exercise Stress:
  * Doses at rest were to range between 1.7 and 2.0 mCi.
  * Doses under stress were to be a factor of 3.0 to 3.6 greater than the rest dose, resulting in a range between 5.1 and 7.2 mCi.
  Other Names: There are no other names

SUMMARY:
The main purpose of this study is to get more information on using BMS747158 (the study drug),a drug with small amounts of radioactivity to allow for heart imaging, during a PET scan which can then be compared to other images such as SPECT. The safety and quality of images will be studied.

DETAILED DESCRIPTION:
The primary objectives of this study are:

* To acquire data for the development of one-day rest/stress cardiac PET perfusion imaging protocols for BMS747158 with comparable diagnostic image quality to a two-day rest/stress PET protocol
* To assess the safety of multiple doses of BMS747158

The secondary objectives of this study are:

* To assess PET imaging parameters and image quality following administration of BMS747158 at rest and at stress (pharmacologic or exercise) same day (at different time intervals) and 16-48 hours after the rest injection
* To assess feasibility of gated cardiac PET imaging with BMS747158 for left ventricular function assessment
* To assess agreement of one and two day rest/stress PET imaging with BMS747158 in patients with reversible ischemia with rest/stress single photon emission computed tomography (SPECT) imaging
* To perform a preliminary assessment of the diagnostic accuracy of one-day and two-day rest/stress PET perfusion imaging with BMS747158 as compared with invasive coronary angiography or computed tomography angiography (CTA) for detection of

ELIGIBILITY:
Inclusion Criteria:

* Provide signed IC prior to undergoing any study procedures
* Be male or nonpregnant female, between the ages of 18 to 75 years, inclusive
* Have:A rest/stress SPECT imaging study (either exercise or pharmacologic stress) within 21 days of enrollment, using 99mTc-labeled tracers and showing reversible ischemia
* Female patients must:

  * be nonlactating,
  * no longer have child-bearing potential, either because they are post-menopausal (defined as amenorrhea ≥ 12 consecutive months, or because they have undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy)

Exclusion Criteria:

* Presence of any condition that may disrupt and/or increase permeability of the BBB, including multiple sclerosis, Alzheimer's disease, Parkinson's disease, acute central nervous system (CNS) infection, CNS tumor, autoimmune disease affecting the CNS, or CNS inflammatory
* Current significant illness, pathology or physical examination or vital signs measurement-findings that could potentiate any adverse pharmacological event associated with a vasodilatory drug or any pathology that, in the opinion of the investigator, might confound the interpretation of the results of the study
* Known hypersensitivity to adenosine, dipyridamole or aminophylline
* Presence of any contraindications to exercise stress testing
* History of New York Heart Association Class III or IV Congestive Heart Failure (CHF)
* Any major surgery within 4 weeks prior to enrollment or planned within 2 weeks following completion of the 2-week telephone follow-up assessment
* Inability to tolerate IV medication.
* History of drug or alcohol abuse within the last year
* Participation in any investigational drug, device, or placebo study within 6 months prior to study enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Orlandi, MD, Study Director — Lantheus Medical Imaging
Locations (24):
- United States (24):
  - Silicon Valley Medical Imaging, Fremont, California
  - Scripps Memorial Hospital, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Medical Plaza, Los Angeles, California
  - Radiological Associates of Sacramento, Sacramento, California
  - VA Healthcare System San Diego, San Diego, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Emory University Hospital, Atlanta, Georgia
  - Primary Care Cardiology Research, Inc, Ayer, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Cardiovascular Consultants, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Columbia University Medical Center, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - University Hospital Case Medical Center, Cleveland, Ohio
  - Midwest Cardiology Research Foundation, Columbus, Ohio
  - Mountain States Health Alliance, Johnson City, Tennessee
  - East Tennessee Clinical Research Institute, Knoxville, Tennessee

REFERENCES:
- [Background] Bateman TM. Cardiac positron emission tomography and the role of adenosine pharmacologic stress. Am J Cardiol. 2004 Jul 22;94(2A):19D-24D; discussion 24D-25D. doi: 10.1016/j.amjcard.2004.04.013. PMID 15261128
- [Background] Beller GA. First annual Mario S. Verani, MD, Memorial lecture: clinical value of myocardial perfusion imaging in coronary artery disease. J Nucl Cardiol. 2003 Sep-Oct;10(5):529-42. doi: 10.1016/s1071-3581(03)00655-x. PMID 14569247
- [Background] Beller GA, Bergmann SR. Myocardial perfusion imaging agents: SPECT and PET. J Nucl Cardiol. 2004 Jan-Feb;11(1):71-86. doi: 10.1016/j.nuclcard.2003.12.002. No abstract available. PMID 14752475
- [Background] Beller GA, Zaret BL. Contributions of nuclear cardiology to diagnosis and prognosis of patients with coronary artery disease. Circulation. 2000 Mar 28;101(12):1465-78. doi: 10.1161/01.cir.101.12.1465. No abstract available. PMID 10736294
- [Background] Cerqueira MD, Verani MS, Schwaiger M, Heo J, Iskandrian AS. Safety profile of adenosine stress perfusion imaging: results from the Adenoscan Multicenter Trial Registry. J Am Coll Cardiol. 1994 Feb;23(2):384-9. doi: 10.1016/0735-1097(94)90424-3. PMID 8294691
- [Background] Guideri F, Ferber D, Galgano G, Isidori S, Blardi P, Pasini FL, Di Perri T. QTc interval prolongation during infusion with dipyridamole or adenosine. Int J Cardiol. 1995 Jan 27;48(1):67-73. doi: 10.1016/0167-5273(94)02209-2. PMID 7744540
- [Background] Glover DK, Gropler RJ. Journey to find the ideal PET flow tracer for clinical use: are we there yet? J Nucl Cardiol. 2007 Nov-Dec;14(6):765-8. doi: 10.1016/j.nuclcard.2007.09.019. No abstract available. PMID 18022101
- [Background] Henzlova MJ, Cerqueira MD, Mahmarian JJ, Yao SS; Quality Assurance Committee of the American Society of Nuclear Cardiology. Stress protocols and tracers. J Nucl Cardiol. 2006 Nov;13(6):e80-90. doi: 10.1016/j.nuclcard.2006.08.011. No abstract available. PMID 17174798
- [Background] Miyamoto MI, Vernotico SL, Majmundar H, Thomas GS. Pharmacologic stress myocardial perfusion imaging: a practical approach. J Nucl Cardiol. 2007 Apr;14(2):250-5. doi: 10.1016/j.nuclcard.2007.01.006. No abstract available. PMID 17386388

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohort 1 enrolled 33 patients across 3 clinical sites. Dosing for Cohort 1 was initiated January 2009.
  Cohort 2 enrolled 143 patients across 21 clinical sites. Dosing for Cohort 2 was initiated July 2009
Pre-assignment Details: Cohort 1: Patients showing a mild to severe reversible perfusion defect on a qualifying SPECT MPI study were considered eligible for the study Cohort 2: Patients with known or suspected cornary artery disease who presented with a broad spectrum of pre-test likelihood of CAD(very low/low, to high likelihood)were considered eligible for the study.
Groups:
- Cohort 1 Dose Ranging and Dose Interval: Patients received 2 or 3 IV bolus injections of BMS747158: 1 at rest and 1 at pharmacologic/exercise stress, over a 1-day or 2-day period
- Cohort 2 Preliminary Efficacy Pharmacologic Stress: Patients received 2 injections of BMS747158: 1 at rest and 1 at Pharmacologic stress, over a 1-day period.
Period: Cohort 1 Dose Ranging and Dose Interval
Arm/Group | Cohort 1 Dose Ranging and Dose Interval | Cohort 2 Preliminary Efficacy Pharmacologic Stress
Started | 33 | 0 (Cohort 2(Pharm Stress) subjects did not participate in dose range, dose frequency)
Completed | 32 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Cohort 2 Efficacy
Arm/Group | Cohort 1 Dose Ranging and Dose Interval | Cohort 2 Preliminary Efficacy Pharmacologic Stress
Started | 0 (Cohort 1 subjects did not participate in period 2: efficacy) | 143
Completed | 0 | 133
Not Completed | 0 | 10
Not completed — Adverse Event | 0 | 1
Not completed — Other | 0 | 9

BASELINE CHARACTERISTICS:
Population: Intent to treat population Cohort 1 N=33; Cohort 2 N=125 Safety population; Cohort 1 N=33; Cohort 2 N=143
Groups:
- Cohort 1 Dose Ranging and Dose Interval: Patients received either 2 or 3 IV bolus injhections of BMS747158: 1 at rest and 1 or 2 during stress, over a 1-day or 2-day period
- Cohort 2: Pharm Stress: Patient received BMS747158 as a single IV bolus injection at rest and a single bolus injection at pharmacologic stress over a 1-day period. For patients undergoing pharmacologic stress test the dose of BMS747158 were to be a factor of 2.0 to 2.4 greater than the rest dose.
- Cohort 2: Efficacy Exercise Stress: Patient received BMS747158 as a single IV bolus injection at rest and a single bolus injection at exercise stress over a 1-day period.
  For patients undergoing exercise stress test the dose of BMS747158 were to be a factor of 3.0 to 3.6 greater than the rest dose.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Dose Ranging and Dose Interval | Cohort 2: Pharm Stress | Cohort 2: Efficacy Exercise Stress | Total
Number analyzed (Participants) | 33 | 67 | 76 | 176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 24 | 52 | 85
  >=65 years | 24 | 43 | 24 | 91
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 20 | 45
  Male | 24 | 51 | 56 | 131
Region of Enrollment [Number; unit: participants]
  North America | 33 | 67 | 76 | 176

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Determination of Rest Dose: Dose Acquistion Time Product
Description: The rest flurpiridaz dose to be used for subsequent efficacy studies was determined by a modeling method that simulated a range of injected doses using a single fixed injected dose at rest in each subject and a range of acquisition durations. From this, a dose acquisition time product (DATP was determined for each subject that specified the minimal dose for a given acquisition duration that yielded an image in that subject that was negligibly affected by photon counting statistics. Descriptive statistics were used to identify an appropriate rest dose for the population. No other statistical tests were performed
Time Frame: Dosing visit
Population: Intent to treat, received at least one rest dose of BMS 747158
Measure: Mean (Standard Deviation); unit: MBq X Minutes
Groups:
- Cohort 1: Dose Acquistion Time Product: Subjects received either 2 or 3 IV bolus injhections of BMS747158: 1 at rest and 1 or 2 during stress, over a 1-day or 2-day period
Arm/Group | Cohort 1: Dose Acquistion Time Product
Number analyzed (Participants) | 33
MBq X Minutes | 100 (54.7)

2. Primary Outcome: Cohort 2: Diagnostic Efficacy of One-day Rest/Stress BMS747158 PET MPI Sensitivity (SN) vs SPECT MPI Sensitivity
Description: Diagnostic efficacy of one-day rest/stress BMS747158 PET MPI is measured by sensitivity as compared to single photon emission computed tomography (SPECT)MPI in the detection of coronary artery disease (CAD)using angiography or three-month cardiac events as the truth standard.
Time Frame: Dosing visit
Population: intent to treat, received at least one dose of BMS747158
Measure: Number; unit: Proportion of True Positive Cases
Groups:
- Cohort 2 Efficacy/Safety: Patient received BMS747158 as a single IV bolus injection at rest and a single bolus injection at stress over a 1-day period. For patients undergoing pharmacologic stress test the dose of BMS747158 were to be a factor of 2.0 to 2.4 greater than the rest dose. For patients undergoing exercise stress test the dose of BMS747158 were to be a factor of 3.0 to 3.6 greater than the rest dose.
Arm/Group | Cohort 2 Efficacy/Safety
Number analyzed (Participants) | 125
Proportion of True Positive Cases
  PET MPI | 0.769
  SPECT MPI | 0.596
Statistical Analysis 1: Comparison: Cohort 2 Efficacy/Safety; Test type: Superiority or Other; p = 0.02, McNemar — P-Value for sensitivity comparison of PET MPI for the same reader; two-sided McNemar test with 1 degree of freedom; sensitivity = 0.769, 95% CI 2-sided [0.655 to 0.884] — No standard deviation can be calculated for PET sensitivity
Statistical Analysis 2: Comparison: Cohort 2 Efficacy/Safety; Test type: Superiority or Other; p = 0.02, McNemar — p-value for sensitivity comparison for SPECT MPI for the same reader; Sensitivity = 0.596, 95% CI 2-sided [0.463 to 0.730] — No standard deviation can be calculated for SPECT sensitivity

3. Primary Outcome: Cohort 1: Determination of Ratio of Stress Dose to Rest Dose
Description: The stress flurpiridaz dose for subsequent same-day rest-stress efficacy studies was determined as a multiple of the rest dose by computer modeling. Images derived only from rest flurpiridaz administration were blended using image analysis with images derived only from administration of flurpiridaz following exercise or adenosine stress. The blending fraction that resulted in negligible change in reader interpretation of defect severity was determined for each subject. The minimum value that met this criterion for all subjects was used to calculate the ratio of the stress dose to the rest dose as a function of the delay between administration of the two doses for both adenosine stress and exercise stress separately. No statistical analysis was performed.
Time Frame: Dosing visit
Population: Subjects with demonstrated partially or completely reversible defects on prior SPECT who received at least one stress and one rest dose of flurpiridaz F 18, on separate days.
Measure: Number; unit: Fraction of rest added to stress image
Groups:
- Cohort 1 Dose Ranging and Dose Interval: Subjects received 2 or 3 IV bolus injections of BMS747158: 1 at rest and 1 at pharmacologic/exercise stress, over a 1-day or 2-day period
Arm/Group | Cohort 1 Dose Ranging and Dose Interval
Number analyzed (Participants) | 26
Fraction of rest added to stress image | 0.228

4. Primary Outcome: Cohort 2: Diagnostic Efficacy of One-day Rest/Stress BMS747158 PET MPI Specificity (SP) vs SPECT MPI Specificity
Description: Diagnostic efficacy of one-day rest/stress BMS747158 PET MPI is measured by specificity as compared to single photon emission computed tomography (SPECT)MPI in the detection of coronary artery disease (CAD)using angiography or three-month cardiac events as the truth standard.
Time Frame: Dosing Visit
Population: intent to treat, received at least one dose of BMS747158
Measure: Number; unit: Proportion of True Negative Cases
Groups:
- Cohort 2: Efficacy/Safety: Patient received BMS747158 as a single IV bolus injection at rest and a single bolus injection at stress over a 1-day period. For patients undergoing pharmacologic stress test the dose of BMS747158 were to be a factor of 2.0 to 2.4 greater than the rest dose. For patients undergoing exercise stress test the dose of BMS747158 were to be a factor of 3.0 to 3.6 greater than the rest dose.
Arm/Group | Cohort 2: Efficacy/Safety
Number analyzed (Participants) | 125
Proportion of True Negative Cases
  PET MPI | 0.877
  SPECT MPI | 0.836
Statistical Analysis 1: Comparison: Cohort 2: Efficacy/Safety; Test type: Superiority or Other; p = 0.317, McNemar — p-value for comparison of PET specificity for same reader; PET specificity = 0.877, 95% CI 2-sided [0.801 to 0.952] — no standard deviation for PET specficity
Statistical Analysis 2: Comparison: Cohort 2: Efficacy/Safety; Test type: Superiority or Other; p = 0.317, McNemar — p-value for comparison of SPECT specificity for same reader; SPECT specificity = 0.836, 95% CI 2-sided [0.751 to 0.921] — no standard deviation for SPECT specificity

ADVERSE EVENTS:
Time Frame: Cohort 1: Adverse event monitoring was initiated on Study Day 1 at time of rest dose and conitnued through 2-week follow up Cohort 2: Adverse event monitoring was intiatied on Study Day 1 at time of rest dose and continued through 1-week follow up
Description: Safety data were not combined and are reported by Cohort
Groups:
- Cohort 1: Dose Range and Dose Interval: Patients to receive either 2 or 3 IV bolus injections of BMS747158: 1 at rest and 1 or 2 during pharmacological or exercise stress, over a 1-day or 2-day period.
  BMS747158: dosages at rest and at stress were not to exceed a total of 14 mCi.
  Cohort 1: Patients received either 2 or 3 IV bolus injections of BMS747158: 1 at rest and 1 or 2 during stress, over a 1-day or 2-day period.
- Cohort 2: Efficacy in Pharm Stress: Patients receive 2 IV injections of BMS747158:at rest and stress
  For the Pharmacologic (Adenosine) Stress:
  * Doses range at rest between 2.9 and 3.4 mCi.
  * Dose range at stress between 5.8 and 8.2 mCi (factor of 2.0 to 2.4 greater than the rest dose).
  For the Exercise Stress:
  * Doses at rest were to range between 1.7 and 2.0 mCi.
  * Doses under stress were to be a factor of 3.0 to 3.6 greater than the rest dose, resulting in a range between 5.1 and 7.2 mCi.
Arm/Group | Cohort 1: Dose Range and Dose Interval | Cohort 2: Efficacy in Pharm Stress
Serious Adverse Events (participants affected / at risk) | 0/33 | 2/143
Other Adverse Events (participants affected / at risk) | 21/33 | 61/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Dose Range and Dose Interval (N=33) | Cohort 2: Efficacy in Pharm Stress (N=143)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Right Knee Effusion
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) — Progressively Worsening Dizziness
Hypertension (Vascular disorders) | 0 (0) | 1 (1) — Progressively worsening Hypertension
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Dose Range and Dose Interval (N=33) | Cohort 2: Efficacy in Pharm Stress (N=143)
Angina Pectoris (Cardiac disorders) | 2 (2) | 6 (6)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 6 (6)
Chest Discomfort (General disorders) | 2 (2) | 9 (9)
Fatigue (General disorders) | 3 (3) | 0 (0)
Feeling Hot (General disorders) | 4 (4) | 0 (0)
INfluenza Like Illness (General disorders) | 1 (1) | 0 (0)
Non Cardiac Chest Pain (General disorders) | 1 (1) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculosketetal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 4 (4)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 10 (10)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 7 (7) | 7 (7)
Claustrophobia (Psychiatric disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days